CLINICAL TRIAL: NCT05368506
Title: An Early Phase I Study of the Pharmacodynamics of WEE1 Inhibitor, ZN-c3, in Metastatic Solid Tumors
Brief Title: ZN-c3 for the Treatment of Metastatic Triple-Negative Breast Cancer and Advanced Ovarian Cancer
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: PI discretion
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Oregon Health and Science University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00022229; NCI-2022-03599 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00022229 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2022-05-05; First posted 2022-05-10 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Advanced Fallopian Tube Carcinoma; Advanced Ovarian Carcinoma; Advanced Primary Peritoneal Carcinoma; Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Triple-Negative Breast Carcinoma; Stage III Fallopian Tube Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Primary Peritoneal Cancer AJCC v8; Stage IV Fallopian Tube Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Primary Peritoneal Cancer AJCC v8
MeSH Terms: conditions — Triple Negative Breast Neoplasms; Fallopian Tube Neoplasms; Ovarian Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (wee1 inhibitor ZN-c3) (Experimental): Patients receive Wee1 inhibitor ZN-c3 PO QD on days 1-21. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: Wee1 Inhibitor ZN-c3

INTERVENTIONS:
Drug: Wee1 Inhibitor ZN-c3 — Given PO
  Other Names: ZN c3; ZN-c3; ZNc3

SUMMARY:
This early phase I trial tests the safety and side effects of ZN-c3 in treating patients with triple-negative breast cancer or ovarian cancer that have spread to other parts of the body (metastatic or advanced). ZN-c3 is an enzyme inhibitor that may stop the growth of cancer cells by blocking some of the enzymes needed for cell growth.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the primary pharmacodynamic effect of wee1 inhibitor ZN-c3 (ZN-c3) in tumor biopsies from patients with advanced triple-negative breast cancer (TNBC) and ovarian cancer.

II. To assess safety and tolerability of the proposed therapy.

SECONDARY OBJECTIVES:

I. To assess clinical benefit of TNBC and ovarian cancer patient from the proposed therapy.

II. To determine time to disease progression. III. To assess participant survival on study.

EXPLORATORY OBJECTIVES:

I. To evaluate ZN-c3 pharmacokinetics (PK). II. To identify predictive biomarkers of sensitivity to therapy. III. To identify emerging mechanisms of resistance to therapy.

OUTLINE:

Patients receive Wee1 inhibitor ZN-c3 orally (PO) once daily (QD) on days 1-21. Treatment repeats every 21 days for up to 12 cycles in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for to 1 year.

ELIGIBILITY:
Inclusion Criteria:

* Participant must provide written informed consent before any study-specific procedures or interventions are performed
* Participants aged >= 18 years
* Participants with biopsy proven metastatic TNBC defined as:

  * Estrogen receptor (ER) < 10%, progesterone receptor (PR) < 10%
  * HER2 non-amplified by College of American Pathologists (CAP) guidelines
* Participants with biopsy proven advanced ovarian cancer (including primary peritoneal and fallopian tube cancers)
* Prior PARP inhibitor therapy allowed
* Participants must have at least one measurable site of disease as defined by Response Evaluation Criteria in Solid Tumors (RECIST) version (v) 1.1 that is amendable to biopsy
* Participants must have received at least one standard of care line of therapy in the recurrent setting
* Eastern Cooperative Oncology Group (ECOG) performance status (PS) =< 2
* Prior treatment related toxicities resolved to =< grade 1 (except neuropathy, alopecia or skin pigmentation)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L; excluding measurements obtained within 7 days after daily administration of filgrastim/sargramostim or within 3 weeks after administration of pegfilgrastim
* Platelet count >= 100 x 10^9/L; excluding measurements obtained within 3 days after transfusion of platelets
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) =< 3 × upper limit of normal (ULN). If liver function abnormalities are due to underlying liver metastases, AST and ALT =< 5 x ULN
* Total serum bilirubin =< 1.5 x ULN or =< 3 x ULN in the case of Gilbert's disease
* Serum creatinine =< 1.5 x ULN or creatinine clearance (CrCl) >= 60 mL/min
* Participants of childbearing potential must have a negative serum beta human chorionic gonadotropin (beta-hCG) test
* Participants of childbearing potential must agree to use an effective method of contraception per institutional standard prior to the first dose and for 90 days after the last dose of ZN-c3
* Willingness and ability to comply with scheduled visits, treatment plan, laboratory tests and other study procedures, including pretreatment and on-treatment biopsies
* Willingness to practice adequate sun protection (use of sunscreen or sun-protective clothing or limitation of sun exposure)

Exclusion Criteria:

* Prior Wee-1 inhibitor exposure
* Any of the following treatment interventions within the specified time frame prior to cycle 1 day 1:

  * Major surgery within 28 days (the surgical incision should be fully healed prior to study drug administration)
  * Radiation therapy within 21 days; however, if the radiation portal covered =< 5% of the bone marrow reserve, the subject is eligible irrespective of the end date of radiotherapy
  * Autologous or allogeneic stem cell transplant within 3 months
  * Current use of an investigational agent that is not expected to be cleared by the first dosing of study drug or that has demonstrated to have prolonged side effects
  * Prescription, non-prescription drugs or food known as moderate to strong inducers of CYP3A within 2 weeks
* A serious illness or medical condition(s) including, but not limited to, the following:

  * Symptomatic brain metastases
  * Leptomeningeal disease that requires or is anticipated to require immediate treatment
  * Myocardial impairment of any cause (e.g., cardiomyopathy, ischemic heart disease, significant valvular dysfunction, hypertensive heart disease, and congestive heart failure) resulting in heart failure by New York Heart Association Criteria (class III or IV)
  * Other severe acute or chronic medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration, or may interfere with the interpretation of study results, and in the judgment of the investigator would make the subject inappropriate for entry into this study
  * Significant gastrointestinal abnormalities, including an inability to take oral medication, requirement for intravenous (IV) alimentation, active peptic ulcer, chronic diarrhea or vomiting considered to be clinically significant in the judgment of the Investigator, or prior surgical procedures affecting absorption
  * Active or uncontrolled infection. Subjects with an infection receiving treatment (antibiotic, antifungal or antiviral treatment) may be entered into the study but must be afebrile and hemodynamically stable for >= 72 hours
* Unresolved toxicity of grade > 1 attributed to any prior therapies (excluding grade 2 neuropathy, alopecia or skin pigmentation)
* Known hypersensitivity to any drugs similar to ZN-c3 in class
* Participants that are pregnant or lactating (including the cessation of lactation) or those of childbearing potential who have a positive serum pregnancy test within 14 days prior to cycle 1 day 1
* Participants with active (uncontrolled, metastatic) second malignancies or requiring therapy
* 12-lead electrocardiogram (ECG) demonstrating a corrected QT interval using Fridericia's formula (QTcF) of > 480 msec, except for subjects with atrioventricular pacemakers or other conditions (e.g., right bundle branch block) that render the QT measurement invalid
* Any history or current evidence of congenital long QT syndrome
* Participant requiring any medications that can lead to significant QT prolongation
* Participant requires administration of strong and moderate CYP3A4 inhibitors and inducers as well as strong and moderate P-glycoprotein (P-gp) inhibitors
* Participants with any condition that, in the opinion of the investigator, could jeopardize the participant's safety or adherence to the study protocol
* For TNBC cohort only, participants with tumors showing androgen receptor (AR) >= 80% by immunohistochemistry are excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-07-30 (Estimated); Primary Completion 2024-09-30 (Estimated); Study Completion 2025-07-31 (Estimated)

PRIMARY OUTCOMES:
Percent decrease of phosphorylated CDK1 and/or Ki67, or p-HH3, or p-CHK1 in tumor cells | Baseline to completion of on-treatment biopsy, up to 21 days
  The point estimate of percentage decrease of either phosphorylated CDK1, or Ki67, or p-HH3, or p-CHK1, or combinations thereof in tumor cells (from baseline) after receiving ZN-c3 will be provided.
Incidence of adverse events | Day 1 to 30 days after last dose of study intervention
  Incidence of grade >= 3 toxicities will be assessed according to Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0.

SECONDARY OUTCOMES:
Clinical benefit rate (CBR) | Day 1 to end of treatment, approximately 12 months
  CBR is the proportion of all participants that achieve a complete response (CR), partial response (PR) or stable disease (SD) >= 6 months without evidence of radiologic progression to this point (i.e., CR + PR + SD)(per Response Evaluation Criteria in Solid Tumors [RECIST] v 1.1).
CBR for ovarian cancer | Day 1 to end of treatment, approximately 12 months
  CBR (i.e., CR + PR + SD) in the ovarian cancer cohort will also be assessed using the Gynecological Cancer Intergroup (GCIG) criteria.
Time to disease progression | Day 1 to date of progression, assessed up to 1 year after discontinuing study drug
  Measure of the length of time from date of study treatment start until the date of cancer progression.
Progression free survival | Day 1 to date of progression or death from any cause, assessed up to 1 year after discontinuing study drug
  Measure of the proportion of participants without disease progression starting from the time from cycle 1 day 1 dose administration to the time of documented disease progression or death from any cause.
Overall survival | Day 1 to death from any cause, assessed up to 1 year after discontinuing study drug
  Measure of the proportion of participants that are alive starting from the time from cycle 1 day 1 dose administration to the time of death from any cause.

OTHER OUTCOMES:
ZN-c3 tumor and plasma concentrations | Baseline to completion of on-treatment biopsy, up to 21 days
  Measure of tumor and plasma concentrations of ZN-c3.
Cellular and molecular characteristics | Baseline to end of study, up to 1 year after discontinuing study drug.
  Descriptive measure of molecular characteristics of patients' tumor

CONTACTS AND LOCATIONS:
Overall Officials: Evthokia Hobbs, M.D., Principal Investigator — OHSU Knight Cancer Institute